CLINICAL TRIAL: NCT05754255
Title: Comparison of High-flow Oxygen With or Without Nasal Positive Airway Pressure (PAP) During Propofol Sedation for Colonoscopy in an Ambulatory Surgical Center: a Prospective Randomized Controlled Trial
Brief Title: Comparison of High-flow Oxygen With or Without Nasal Positive Airway Pressure (PAP) During Propofol Sedation for Colonoscopy in an Ambulatory Surgical Center
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No available resources.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17675
Record Dates: First submitted 2022-12-31; First posted 2023-03-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Colonoscopy; Positive-Pressure Respiration
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A: standard care with a nasal cannula. (Active Comparator): Group A will be given the standard nasal cannula during sedation. The cannula prongs will be inserted into the patient's nose to provide oxygen to the patient.
  Interventions: Device: Nasal Cannula
- Group B: SuperNO2VA™EtCO2 (Active Comparator): Group B will be given a nasal oxygen to deliver gas, create a seal, and provide positive pressure. The mask will be placed over a patient's nose and connected to either an anesthesia circuit or hyperinflation bag during respiratory, anesthesia, and resuscitation procedures.
  Interventions: Device: Nasal Positive Airway Pressure System

INTERVENTIONS:
Device: Nasal Cannula — A nasal cannula is a medical device to provide supplemental oxygen therapy to people who have lower oxygen levels. There are two types of nasal cannulas: low flow and high flow.
  The device has two prongs and sits below the nose. The two prongs deliver oxygen directly into your nostrils.
  Arms: Group A: standard care with a nasal cannula.
Device: Nasal Positive Airway Pressure System — Positive airway pressure (PAP) treatment uses a machine to pump air under pressure into the airway of the lungs. This helps keep the windpipe open during sleep. The forced air delivered by CPAP (continuous positive airway pressure) prevents episodes of airway collapse that block the breathing in people with obstructive sleep apnea and other breathing problems.
  Other Names: Nasal CPAP
  Arms: Group B: SuperNO2VA™EtCO2

SUMMARY:
The primary objective of the prospective study is to compare the incidence, duration, and severity of oxygen desaturation in high-risk patients randomized to nasal mask with nasal positive airway pressure (PAP) or standard care (nasal cannula) receiving propofol sedation during colonoscopy in an ambulatory surgical center (ASC).

Patients will be randomized in groups of ten to one of two groups using a random number table.

Group A: standard care with a nasal cannula. Group B: SuperNO2VA™EtCO2. Following the procedure subjects will be asked to complete satisfaction surveys before leaving the ASC and 48 +/- hours following their procedure.

Researchers will compare levels of satisfaction and levels of oxygen saturation.

DETAILED DESCRIPTION:
This study involves the oxygenation, continuous positive airway pressure, and ventilation of a subject via nasal mask and oxygenation via a closed facemask. The interventions directly related to this study are that of supplement oxygen, bag-mask ventilation, and continuous nasal CPAP intra-operatively and in the recovery unit.

Patients will be randomized in groups of ten to one of two groups using a random number table.

Group A: standard care with a nasal cannula. Group B: SuperNO2VA™EtCO2. For each anesthetic case, a preoperative history and physical and intraoperative record will be documented.

Once in the endoscopy suite, the patients will have baseline vital signs, EtCO2 and oxygen levels measured. Continuous monitoring of heart rate, end tidal CO2 (EtC02), O2 saturation, and every 3-minutes BP monitoring will be obtained. For patients randomized to group A, the anesthesia provider will supply oxygen via nasal cannula at 10LPM. For patients randomized to group B, the anesthesia provider will attach the SuperNO2VA™ EtCO2's circuit port to the hyperinflation bag with the oxygen flow rate to 10 L/min, and the adjustable pressure-limiting (APL) valve completely closed. Initial propofol bolus of 0.5-1.0 mg/kg actual body weight will be administered for sedation. No other sedative or analgesic will be permitted besides propofol. MOAA/S scores will be assessed by the anesthesiologist and medical team and recorded by the research assistant. If the patient's MOAA/S score is ≥ 4, additional 20-50 mg boluses will be administered every 30 - 90 seconds until a MOAA/S score <4 is reached. Once a MOAA/S <4 is reached the endoscopist will insert the colonoscope into the rectum. Sedation will be titrated to maintain a MOAA/S <4 throughout the procedure. If the patient's MOAA/S score ≥4, additional 20-50 mg boluses of propofol will be administered every 30-90 seconds until the MOAA/S is <4. The measurements recorded during colonoscopy for both groups will be: time of administration of sedation; incidence, severity, and duration of oxygen desaturation; number, duration and reason for performing the airway maneuver(s); duration of the procedure; total dose of medication; blood pressure, heart and respiratory rate, and oxygen saturation; time to full recovery; and patient cooperation. The research assistant will document their patient's depth of sedation, cooperation with procedure, and safety.

Endoscope techniques performed during the procedure such as biopsies, dilation, polypectomy, etc. will be tracked. Techniques to facilitate proximal passage of the endoscope such as moving the patient or abdominal pressure will also be noted. If the anatomic extent desired to complete the colonoscopy is not reached (i.e., colon stricture, excessive looping of the instrument), then the patient will be withdrawn from the study.

Patients will recover in the endoscopy suite. The patients will have continuous monitoring of heart rate, end tidal CO2 (EtC02), O2 saturation, and every 5-minute BP monitoring and MOAAS Score. Once a MOAAS score of 5 is obtained, the patient will be offered to drink independently unless deemed inappropriate by the treating physician(s). The endoscopist when available will discuss findings with the patient and/or family, the patient will then dress and leave the endoscopy suite when possible. The time to discharge will be obtained for each patient. Patients will also complete a satisfaction and pain questionnaire before discharge. Subjects will be sent surveys to complete at 48 hours post discharge, concerning their satisfaction and their subjective degree of impairment due to the sedation. They will have the option to complete this electronically via a link to REDCap or with a self-addressed envelope and paper form of the survey. If the patients do not complete or send back their questionnaire, someone will contact them by telephone to collect the data. A statistician using student T-test, Fishers exact test, and other statistical methods they deem appropriate will analyze the collected data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Outpatients undergoing colonoscopy.
3. American Society of Anesthesiology (ASA) Physical Status I-III
4. BMI ≥35 kg/m2, documented obstructive sleep apnea or BMI>30 with STOP-BANG score ≥3
5. Written informed consent

Exclusion Criteria:

1. Inpatient status
2. Active Congestive Heart Failure Exacerbation
3. Untreated ischemic heart disease
4. Acute exacerbation of respiratory disorders, including COPD and asthma
5. Emergent procedures
6. Pregnancy
7. Previous enrollment in this study
8. Inability to provide informed consent.
9. Additional medical testing planned for the same day.
10. History of allergic reaction to propofol
11. History of allergic reaction to polypropylene or PVC.
12. Tracheostomy
13. Supra-glottic or sub-glottic tumor
14. Gastrointestinal tract obstruction or delayed transit (including delayed gastric emptying, gastric bezoar, achalasia, toxic megacolon).
15. Known obstructing colon tumor, lesion, or stricture
16. Previous colon surgery (excluding anal surgery)
17. Active GI bleeding (hematochezia or melena during procedure preparation)
18. Large polyp (> 2cm) removal
19. Previous failed or unsuccessfully completed colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of desaturation | 60 minutes
  Compare incidence of desaturation of Nasal PAP Versus Nasal Administration of Oxygen
Duration of oxygen desaturation | 60 minutes
  Compare the duration of desaturation of Nasal PAP Versus Nasal Administration of Oxygen
Severity of oxygen desaturation | 60 minutes
  Compare the severity of desaturation of Nasal PAP Versus Nasal Administration of Oxygen

SECONDARY OUTCOMES:
Total Amount of Propofol for Adequate Sedation | 60 minutes
  Compares amounts of Propofol for induction and entire procedure administered for procedure
Modified Observer's Assessment of Alertness/Sedation Scale | 60 minutes
  Compare Modified Observer's Assessment of Alertness/Sedation Scale (MOAAS) scores immediately prior to endoscope insertion and during the procedure.
  MOAAS scale is 0-5, where 0=No response after painful stimuli and 5 Responds to name spoken in normal tone. Patients with a MOAAS <4 are considered to be moderately to deeply sedated. The greater the degree of sedation the greater the degree of respiratory depression.
Endoscope Insertion | 60 minutes
  Compare the length of time from induction to endoscope insertion.
Incidence of Airway maneuvers | 60 minutes
  Compare the number of incidence of airway maneuvers
Duration of Airway maneuvers | 60 minutes
  Compare the duration for airway maneuvers
Patient Satisfaction | 48 hours
  Compare patient satisfaction scores (visual analog scale (VAS)) immediately after procedure.
  VAS range is from 0= Not at all satisfied to 5=Completely satisfied.
Reason(s) for airway maneuvers | 60 minutes
  Compare reason(s) for airway maneuvers as reported by anesthesiologist via open ended interview in real time.
Incidence of any desaturation | 60 Minutes
  Compare the incidence of any oxygen desaturation <85% between the start and end of sedation.
Frequency of Oxygen Saturation | 60 minutes
  Compare the frequency of oxygen saturation saturation <85% over 15 seconds between the start and end of sedation.
Frequency of bradycardia | 60 minutes
  Compare the frequency of bradycardia (HR<45 bpm)between the start and end of sedation.
Frequency of low respiratory rate | 60 minutes
  Compare the frequency of low respiratory rate (<6 per minute between the start and end of sedation.
Use of endotracheal intubation | 60 minutes
  Compare the use of endotracheal intubation as airway management in patient population.
Use of Noninvasive positive pressure ventilation | 60 minutes.
  Compare the use of noninvasive positive pressure ventilation as airway management in patient population during sedation.
Use of pharmacological blood pressure support | 60 minutes.
  Compare the use of pharmacological blood pressure support from the start and end of sedation.
Incidence of hospitilization | 48 hours
  Compare the incidence of hospitalization following sedation for a colonoscopy in patient population.
Serious Adverse Events | 48 hours
  Compare incidence of adverse events from start of sedation to 48 hours following the end of sedation.
Frequency of Procedural Interruption | 60 minutes
  Compare the frequency of the removal of endoscope due to a respiratory complication from start to end of sedation.
Duration of Procedural Interruption | 60 minutes.
  Compare the duration of endoscope removal due to a respiratory complication from start of sedation to end of sedation.
Length of Procedure | 60 minutes
  Compare the length of time for procedure from start of sedation to end of sedation.
Ready to discharge | 30 min
  Compare the length of time from end of sedation to ready to discharge
Time to discharge | 90 minutes
  Compare the length of time from end of sedation to actual discharge.

CONTACTS AND LOCATIONS:
Overall Officials: John DeWitt, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States